CLINICAL TRIAL: NCT06841692
Title: Diuretic Testing in Chronic Kidney Disease
Acronym: U-TUBE 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: European Research Council (Other)
Responsible Party: Principal Investigator, Ewout Hoorn, Prof.dr. E.J. Hoorn, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MEC-2024-0799; 101125504 (Other Grant/Funding Number: European Research Council); NL-005327 (Other: Onderzoeksportaal); NL87576.078.24 (Other: Toetsing Online)
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Kidney Disease, Chronic
Keywords: Disease Progression; Diuretic Testing; Chronic Kidney Disease; Kidney Tubular Function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diuretic Group (Experimental): Administration of diuretics on the test day
  Interventions: Diagnostic Test: Diuretic Testing
- Time control group (No Intervention): No diuretics will be administered

INTERVENTIONS:
Diagnostic Test: Diuretic Testing — The administration of hydrochlorothiazide and bumetanide is used to stimulate and assess tubular function.
  Arms: Diuretic Group

SUMMARY:
The goal of this clinical trial is to predict the progression of chronic kidney disease by diuretic testing in patients with chronic kidney disease. The main questions it aims to answer are:

Does a worse result of a diuretic test predict the progression of chronic kidney disease?

If there is a comparison group: Researchers will compare the diuretic test in patients with chronic kidney disease to healthy participants to see if the results are different in a healthy kidney.

Participants will undergo diuretic testing. This involves the administration of bumetanide and hydrochlorothiazide with subsequent blood and urine collections.

ELIGIBILITY:
Inclusion Criteria for CKD subjects:

* CKD stage G3 (creatinine-based eGFR 30-59 mL/min/1.73m2) during the last outpatient visit

Inclusion Criteria for Healthy subjects:

• eGFR within the expected range for age (a decline of 1 ml/min/1.73 m2 per year starting from age 40 is considered the normal age-related decline in kidney function

Exclusion Criteria:

* Known intolerance or allergy to the diuretics
* Current systemic chemotherapy for malignancy
* Kidney transplant recipient
* Use of calcineurin-inhibitors
* Life expectancy < 12 months
* Current immunosuppressive treatment for glomerulonephritis
* Incapacitated subjects or subjects who are deemed unfit to adequately adhere to instructions from the research team
* Hypokalemia or hyperkalemia (K+ < 3.0mmol/L or K+ > 5.5 mmol/L) at inclusion visit
* Hypo- or hypernatremia (Na+ < 130 mmol/L or Na+ > 150mmol/L) at inclusion visit
* Inherited tubulopathy as the cause of CKD
* Autosomal dominant polycystic or tubulointerstitial kidney disease causing CKD
* Clinically relevant heart failure (New York Heart Association class III or IV)
* Therapy-resistant hypertension, defined as systolic blood pressure > 180mmHg at the inclusion visit
* Current treatment with inhibitors of Organic anion transporters: probenecid, pravastatin, cimetidine, cephalosporins, acetazolamide [22]
* Active hepatitis during last outpatient visit
* Liver cirrhosis in advanced stage (Child-Pugh B or C)
* Active drug- or alcohol abuse
* Not being able to tolerate a 28-day washout of one of the drugs interfering with diuretic testing.
* Women who are pregnant, breastfeeding, or planning on becoming pregnant before the test day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression of Chronic Kidney Disease | 3 years
  This composite outcome consists of the reduction of kidney function of 30% measured as creatinine-based estimated glomerular filtration rate (eGFR) using the chronic kidney disease epidemiology collaboration (CKD-EPI) 2021 formula or the initiation of kidney replacement therapy (dialysis or kidney transplantation)

CONTACTS AND LOCATIONS:
Overall Officials: Ewout J. Hoorn, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colussi G, Bettinelli A, Tedeschi S, De Ferrari ME, Syren ML, Borsa N, Mattiello C, Casari G, Bianchetti MG. A thiazide test for the diagnosis of renal tubular hypokalemic disorders. Clin J Am Soc Nephrol. 2007 May;2(3):454-60. doi: 10.2215/CJN.02950906. Epub 2007 Mar 14. PMID 17699451
- [Background] Chawla LS, Davison DL, Brasha-Mitchell E, Koyner JL, Arthur JM, Shaw AD, Tumlin JA, Trevino SA, Kimmel PL, Seneff MG. Development and standardization of a furosemide stress test to predict the severity of acute kidney injury. Crit Care. 2013 Sep 20;17(5):R207. doi: 10.1186/cc13015. PMID 24053972
- [Background] Rodriguez-Iturbe B, Herrera J, Marin C, Manalich R. Tubular stress test detects subclinical reduction in renal functioning mass. Kidney Int. 2001 Mar;59(3):1094-102. doi: 10.1046/j.1523-1755.2001.0590031094.x. PMID 11231365